CLINICAL TRIAL: NCT03889210
Title: Cross-over, Placebo-controlled, Randomized Trial of β-hydroxybutyrate in Prediabetes
Brief Title: β-hydroxybutyrate, Glucose Metabolism and Prediabetes
Acronym: CETUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Max Petrov, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 18/NTB/161
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: PreDiabetes
Keywords: Ketones; Prediabetes
MeSH Terms: conditions — Prediabetic State; Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HVMN ketone drink (Active Comparator): HVMN ketone drink will be given in a total volume of 100 ml.
  Interventions: Other: HVMN Ketone
- Placebo (Placebo Comparator): Placebo will be given in a total volume of 100 ml.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: HVMN Ketone — Water-based, flavoured sport beverage
  Arms: HVMN ketone drink
Other: Placebo — Water, stevia, malic acid, and thickening agent
  Arms: Placebo

SUMMARY:
The study aims to investigate changes in blood glucose metabolism after administration of a ketone ester drink.

DETAILED DESCRIPTION:
New-onset prediabetes is the most significant risk factor for diabetes. Clinical studies in healthy human volunteers have demonstrated that ketone esters lower blood glucose levels in both fasting and fed state.

Participants will visit the COSMOS clinic on two occasions and will be randomly allocated to receive either the HVMN ketone drink or placebo, in a cross-over design. Blood samples will be collected sequentially every 30 minutes for up to 150 minutes. Blood samples will be assayed for glucose and other markers of glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over 18 years
* Individuals diagnosed with prediabetes; defined based on the American Diabetes Association guidelines
* History of at least one episode of acute pancreatitis
* Written informed consent

Exclusion Criteria:

* Individuals who are on a ketogenic diet or consuming nutritional ketone supplements
* History of cancer or chronic pancreatitis
* History of bariatric or gastrointestinal surgery
* Pregnant or breastfeeding women
* Individuals involved in intensive endurance training or competitive athletics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Rate of change in plasma glucose concentration | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma glucose concentration before and after administration of the intervention/placebo

SECONDARY OUTCOMES:
Rate of change in plasma insulin and C-peptide concentrations | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma insulin and C-peptide concentrations before and after administration of the intervention/placebo
Rate of change in plasma concentration of gut and pancreatic hormones | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma concentrations of ghrelin, incretins, cholecystokinin, gastrin-releasing peptide, peptide YY, oxyntomodulin, motilin, glucagon, amylin, pancreatic polypeptide, and vasoactive intestinal peptide before and after administration of the intervention/placebo
Rate of change in lipid profile and digestive enzymes | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma concentration of triglycerides, glycerol, cholesterol, lipases before and after administration of the intervention/placebo
Rate of change in plasma concentration of pro-inflammatory cytokines | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma concentration of interleukin-1β, interleukin-6, leptin, tumor necrosis factor α, and monocyte chemoattractant protein-1 and other cytokines before and after administration of the intervention/placebo
Rate of change in plasma concentration of markers of iron metabolism | Baseline, 30, 60, 90, 120, and 150 minutes
  Changes in plasma concentration of ferritin, hepcidin, transferrin receptor before and after administration of the intervention/placebo
Correlation with body fat phenotypes | 150 minutes
  Differences in the association between rate of change in plasma glucose concentration and magnetic resonance imaging-derived visceral fat volume in the intervention/placebo
Correlation with body fat phenotypes | 150 minutes
  Differences in the association between rate of change in plasma glucose concentration and magnetic resonance imaging-derived subcutaneous fat volume in the intervention/placebo
Correlation with body fat phenotypes | 150 minutes
  Differences in the association between rate of change in plasma glucose concentration and magnetic resonance imaging-derived liver fat per centage in the intervention/placebo
Correlation with physical activity | 150 minutes
  Differences in the association between rate of change in plasma glucose concentration and metabolic equivalents score in the intervention/placebo

CONTACTS AND LOCATIONS:
Locations (1):
- University of Auckland; Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Charles S, Liu Y, Bharmal SH, Kimita W, Petrov MS. Effect of Acute Nutritional Ketosis on Circulating Levels of Growth Differentiation Factor 15: Findings from a Cross-Over Randomised Controlled Trial. Biomolecules. 2024 Jun 6;14(6):665. doi: 10.3390/biom14060665. PMID 38927068
- [Derived] Charles S, Liu Y, Kimita W, Ko J, Bharmal SH, Petrov MS. Effect of D-beta-hydroxybutyrate-(R)-1,3 butanediol on plasma levels of asprosin and leptin: results from a randomised controlled trial. Food Funct. 2023 Jan 23;14(2):759-768. doi: 10.1039/d2fo02405e. PMID 36594212
- [Derived] Liu Y, Bharmal SH, Kimita W, Petrov MS. Effect of d-beta-Hydroxybutyrate-(R)-1,3 Butanediol on Appetite Regulation in People with Prediabetes. Mol Nutr Food Res. 2023 Feb;67(4):e2200615. doi: 10.1002/mnfr.202200615. Epub 2023 Jan 26. PMID 36565045
- [Derived] Liu Y, Bharmal SH, Kimita W, Petrov MS. Effect of acute ketosis on lipid profile in prediabetes: findings from a cross-over randomized controlled trial. Cardiovasc Diabetol. 2022 Jul 23;21(1):138. doi: 10.1186/s12933-022-01571-z. PMID 35871064
- [Derived] Bharmal SH, Alarcon Ramos GC, Ko J, Petrov MS. Abdominal fat distribution modulates the metabolic effects of exogenous ketones in individuals with new-onset prediabetes after acute pancreatitis: Results from a randomized placebo-controlled trial. Clin Nutr ESPEN. 2021 Jun;43:117-129. doi: 10.1016/j.clnesp.2021.03.013. Epub 2021 Mar 21. PMID 34024503
- [Derived] Bharmal SH, Cho J, Alarcon Ramos GC, Ko J, Cameron-Smith D, Petrov MS. Acute Nutritional Ketosis and Its Implications for Plasma Glucose and Glucoregulatory Peptides in Adults with Prediabetes: A Crossover Placebo-Controlled Randomized Trial. J Nutr. 2021 Apr 8;151(4):921-929. doi: 10.1093/jn/nxaa417. PMID 33561274